CLINICAL TRIAL: NCT07264166
Title: Healing Hope International Multinational Observational Registry Evaluating Intranasal 15-Gene AAV9-PHP.eB Therapy and Functional Outcomes in Children With Chronic Hypoxic-Ischemic Encephalopathy (GEN-HOPE Study)
Brief Title: International Observational Study of Intranasal 15-Gene AAV9-PHP.eB Therapy for Children With Chronic Hypoxic-Ischemic Encephalopathy (Cerebral Palsy)
Acronym: GEN-HOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Healing Hope International (Other)
Responsible Party: Principal Investigator, Tamara C Tamas, Director of Clinical Research, Healing Hope International
Other Study IDs: HHI-HIE-OBS-2025-001
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hypoxic Brain Damage; Hypoxic Ischaemic Encephalopathy (HIE); Hypoxic Ischaemic Encephalopathy Due to Cardiac Arrest; Hypoxic Ischemic Encephalopathy of Newborn; Cerebral Palsy; Cerebral Palsy (CP); Cerebral Palsy Hemiparetic Cerebral Palsy Spasticity Gait Disorders, Neurologic Postural Balance Impairment; Cerebral Palsy Quadriplegic; Cerebral Palsy Spastic Diplegia
Keywords: Hypoxic-Ischemic Encephalopathy; HIE; Cerebral Palsy
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia-Ischemia, Brain; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intranasal 15-Gene AAV9-PHP.eB Therapy Cohort: This cohort includes children diagnosed with chronic hypoxic-ischemic encephalopathy (HIE) who receive an intranasal 15-gene AAV9-PHP.eB therapy as part of their existing medical care at participating international sites.

SUMMARY:
This international study, organized by Healing Hope International, is an observational registry designed to collect real-world data on children living with chronic hypoxic-ischemic encephalopathy (HIE) who receive an emerging intranasal gene therapy based on the AAV9-PHP.eB viral vector.

The investigational therapy delivers a panel of 15 restorative genes that support brain repair, reduce inflammation, promote myelination, and improve neural communication. It is administered intranasally in one or three sessions by participating international clinical teams. Because the therapy is already being offered abroad, this registry does not assign treatment but instead follows children who have received it as part of their existing medical care.

The GEN-HOPE Study aims to understand how this gene therapy affects movement, cognition, spasticity, and seizure frequency over time. Families and clinicians will share outcomes such as changes in gross motor function (GMFM-66/88), cognitive assessments (Bayley or WISC tests), and quality-of-life measures. Information on safety, laboratory results, MRI findings, and caregiver-reported experiences will also be collected.

By combining data from multiple countries, the registry seeks to evaluate whether this novel gene-based approach can meaningfully improve daily function and comfort for children with chronic HIE. Results will guide future clinical-trial development and help define safe and effective standards of care for regenerative neurologic therapies.

DETAILED DESCRIPTION:
The GEN-HOPE Study is a multinational, real-world observational registry coordinated by Healing Hope International to evaluate the safety and functional outcomes of a 15-gene AAV9-PHP.eB intranasal gene therapy administered to children with chronic hypoxic-ischemic encephalopathy (HIE) outside the United States.

This registry does not assign or direct any medical intervention. Instead, it prospectively collects standardized clinical and caregiver-reported data from participating international sites where the therapy is already being used under local medical supervision. The aim is to document the naturalistic course of recovery following treatment and to generate evidence that may inform the design of future controlled trials.

The investigational therapy uses an AAV9-PHP.eB viral vector optimized for central nervous system delivery through the nasal mucosa. The 15-gene panel encodes factors related to neuronal plasticity, white-matter repair, anti-inflammatory modulation, metabolic and vascular support, and cellular longevity. Dosing schedules vary by site (single-session or three-session delivery), and some centers administer short-term rapamycin as an adjunctive immunomodulator.

Participants are children aged 2-65 years who have documented chronic HIE, stable baseline medical status, and caregiver consent to share outcome data. Key assessments include gross motor function (GMFM-66/88), cognitive and language evaluations (Bayley-III/IV or WISC-V), spasticity and seizure frequency, and quality-of-life and caregiver burden metrics. Whenever available, MRI/DTI data and laboratory monitoring are recorded. Follow-up intervals occur at approximately 3, 6, 12, 18, and 24 months post-treatment.

Data are analyzed using target-trial emulation and propensity-weighted methods to estimate treatment effects compared with matched external controls receiving standard care. The primary outcome is change in GMFM-66/88 score at 12 months. Secondary outcomes include cognitive performance, seizure burden, quality of life, and safety parameters.

All information is de-identified and stored in a secure international database compliant with data-protection and ethical-governance standards. Oversight is provided by an independent Data and Safety Monitoring Board (DSMB) with expertise in pediatric neurology, statistics, and gene-therapy safety.

The GEN-HOPE Study seeks to accelerate understanding of gene-based neurorestorative strategies and to establish a transparent evidence base supporting compassionate-use access, long-term safety monitoring, and eventual clinical-trial harmonization for children affected by HIE worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 to 65 years, at the time of enrollment.
2. Documented diagnosis of chronic hypoxic-ischemic encephalopathy (HIE), confirmed by medical history, MRI findings, or neonatal records.
3. Stable medical condition for at least 6 months prior to enrollment (no major surgeries or hospitalizations related to HIE within that period).
4. Baseline Gross Motor Function Measure (GMFM-66 or GMFM-88) score between 40% and 70%, representing moderate functional impairment.
5. Completion or active receipt of intranasal 15-gene AAV9-PHP.eB therapy at a participating international clinical site under local physician supervision.
6. Parent(s) or legal guardian(s) willing and able to provide written informed consent for participation in the observational registry and data sharing.
7. Access to clinical follow-up and ability to participate in scheduled assessments or data submissions at 3, 6, 12, 18, and 24 months after treatment.

Exclusion Criteria:

1. Active systemic infection, immune deficiency, or ongoing use of immunosuppressive agents (other than short-term rapamycin used per treating physician's protocol).
2. Known positive anti-AAV9 neutralizing antibody titer at baseline exceeding threshold values that may preclude effective vector transduction (if testing performed locally).
3. Uncontrolled seizure activity exceeding five episodes per day at baseline despite medical therapy.
4. Known or suspected malignancy, severe hepatic or renal dysfunction, or other conditions that would confound safety monitoring.
5. Previous gene therapy or investigational stem cell therapy within the past 12 months.
6. Known pregnancy or breastfeeding in post-pubertal female participants.
7. Any condition that, in the opinion of the local investigator or registry sponsor, may interfere with participation, data reliability, or patient safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients aged 2 to 60 years with chronic hypoxic-ischemic encephalopathy (HIE) who have undergone or are undergoing intranasal 15-gene AAV9-PHP.eB gene therapy at participating international clinical sites.
  Participants typically present with moderate to severe motor and cognitive impairments resulting from neonatal brain injury. Most rely on rehabilitative therapies such as occupational, physical, or speech therapy, and many have comorbid spasticity, seizure disorders, or feeding and respiratory challenges.
  Families voluntarily enroll to share functional, cognitive, imaging, and quality-of-life outcomes following the therapy, allowing the registry to capture real-world data from diverse treatment centers. Enrollment is open to patients meeting medical stability criteria and caregiver consent requirements, regardless of geographic origin, socioeconomic background, or previous therapy history.
  No healthy volunteers are included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM-66/88) Score From Baseline to 12 Months | Baseline to 12 months after treatment
  Assesses change in overall motor ability using the Gross Motor Function Measure (GMFM-66/88), a validated scale for children with cerebral palsy and hypoxic-ischemic injury. Measures performance in lying, sitting, crawling, standing, and walking domains. Higher scores indicate greater motor function.

SECONDARY OUTCOMES:
Change in Cognitive Performance Score | Baseline to 12 months and 24 months
  Evaluated using age-appropriate standardized assessments: Bayley Scales of Infant and Toddler Development (Bayley-III/IV) for ages 2-4, and Wechsler Intelligence Scale for Children (WISC-V) for ages 5-10. Higher scores reflect improved cognitive and developmental performance.
Change in Seizure Frequency | Baseline to 12 months and 24 months
  Monthly caregiver-reported seizure logs and medication records are collected to quantify changes in seizure frequency. Reduction in seizure rate indicates improvement in neuronal stability and anti-inflammatory response.
Change in Spasticity Using the Modified Ashworth Scale (MAS) | Baseline to 12 months
  Measures tone and resistance in major muscle groups using the Modified Ashworth Scale (0 = no increase in tone; 4 = rigid in flexion or extension). Lower scores indicate reduced spasticity.
Change in Quality of Life (PedsQL Caregiver-Reported Score) | Baseline to 12 months and 24 months
  Assesses child and caregiver quality of life using the Pediatric Quality of Life Inventory (PedsQL). Higher scores represent improved perceived quality of life.
Change in MRI/DTI Biomarkers of White-Matter Integrity | Baseline to 12 months
  Quantitative analysis of fractional anisotropy and mean diffusivity from diffusion tensor imaging (DTI) in periventricular and cortical regions. Increases in fractional anisotropy and cortical thickness suggest structural neurorepair.

OTHER OUTCOMES:
Change in Caregiver Burden Score | Baseline to 12 months and 24 months
  Measured using the Caregiver Strain Index (CSI). Lower scores indicate reduced physical, emotional, and time-related burden associated with caregiving.
Incidence of Adverse Events and Serious Adverse Events | Treatment through 24-month follow-up
  Safety endpoints include frequency and severity of adverse events, infections, seizure exacerbations, or hospitalization following gene therapy administration.
Change in Functional Communication (PEDI-CAT / CP-CHILD) | Baseline to 12 months
  Evaluates communication and social interaction using validated scales (PEDI-CAT Communication Domain and CP-CHILD). Higher scores indicate improved communication function.
Change in Laboratory Safety Parameters During Rapamycin Use | Baseline, Weeks 2, 4, 8, and 12
  Monitors complete blood count, liver enzymes, renal profile, and lipid panel in participants receiving adjunctive rapamycin.
Change in Anti-AAV9-PHP.eB Antibody Titers | Baseline to 6 months post-treatment
  Quantifies humoral immune response to AAV9-PHP.eB using ELISA or equivalent assays where available.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anna Lara Kattan, MD: Regenerative Medicine, Principal Investigator — Stem Solutions
Locations (1):
- Stem Solutions, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be publicly shared because the registry collects information from medically fragile children with hypoxic-ischemic encephalopathy across international sites. The data contain potentially identifiable clinical and imaging information that cannot be fully anonymized without risk of re-identification.
  De-identified, aggregate-level results and statistical summaries will be made available through peer-reviewed publications, conference presentations, and registry updates. Access to limited, de-identified datasets for qualified researchers may be considered under controlled data-use agreements and ethics committee approval.

REFERENCES:
- [Background] Lindvall O, Bjorklund A. Cell replacement therapy: helping the brain to repair itself. NeuroRx. 2004 Oct;1(4):379-81. doi: 10.1602/neurorx.1.4.379. No abstract available. PMID 15717041
- [Background] Douglas-Escobar M, Weiss MD. Hypoxic-ischemic encephalopathy: a review for the clinician. JAMA Pediatr. 2015 Apr;169(4):397-403. doi: 10.1001/jamapediatrics.2014.3269. PMID 25685948